CLINICAL TRIAL: NCT05953363
Title: Multi-center, Prospective, Open Label, Single Arm Post-market Study of BD NRFit™ Spinal Needles, NRFit™ Spinal Introducer Needles, and NRFit™ Syringes on Participants Who Are Receiving Neuraxial Procedure.
Brief Title: Prospective Clinical Evaluation of BD NRFit™ Devices and Accessories.
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: MDS-21NRFit001
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Participants who require a BD NRFit™ Spinal Needles, NRFit™ Spinal Introducer Needles, and NRFit™ Syringes as part of their routine medical care.
  Interventions: Device: BD NRFit™ Spinal Needles, BD NRFit™ Spinal Introducer Needles, and BD NRFit™ Syringes

INTERVENTIONS:
Device: BD NRFit™ Spinal Needles, BD NRFit™ Spinal Introducer Needles, and BD NRFit™ Syringes — Insertion of a BD NRFit™ spinal needle and optional BD NRFit™ Spinal Introducer Needle using a BD NRFit™ Syringe to perform the neuraxial procedure.

SUMMARY:
Multi-center, prospective, open label, single arm post-market study to assess the real-world safety and efficacy of BD NRFit™ Spinal Needles, BD NRFit™ Spinal Introducer Needles, and BD NRFit™ Syringes used in an on-market fashion.

DETAILED DESCRIPTION:
This is a multi-center, prospective, open label, single arm post-market study that will enroll approximately 180 participants in order to have a minimum of 150 treated participants who will receive a spinal anesthesia procedure as part of their routine medical care. Participants will be followed from the time of enrollment for up to 10 days (± 3 days) post spinal anesthesia procedure for evidence of adverse events including Post Dural Puncture Headache (PDPH). This can be done via phone if the participant is discharged from the hospital. The site staff must take advantage of the time window of ± 3 days only when the 10-day post-procedure occurs during the weekends or holidays. Any adverse event or complication must be diagnosed and confirmed by a study physician.

A minimum of 50 participants for each of the two needle tip types (Quincke and Whitacre tip) will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient, regardless of age or gender, for which the investigator has decided that a neuraxial procedure must be performed utilizing BD NRFit™ Spinal Needles, NRFit™ Spinal Introducer Needles, and NRFit™ Syringes as part of their routine medical care.
2. Expected to be available for observation through the study period (10 days, ± 3 days, post procedure*).
3. Able and willing to provide signed and dated informed consent or legal authorized representative (LAR) authorized to give consent on behalf of the participant (Note: Consent of guardian or parent may be required for participants under the age of 18 years; participant assent may be required as well).

Exclusion Criteria:

1. Coagulopathy or bleeding disorder, where it is in the opinion of the investigator makes regional anesthetic of increased risk.
2. Subjects with a history of neurological impairment of the trunk or lower extremities.
3. Infection at the site of needle insertion.
4. Previous spine surgery at the level involved in the study procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who will receive a spinal anesthesia procedure as part of their routine medical care.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Hoerauf, MD, Study Director — Becton, Dickinson and Company
Locations (5):
- Austria (2):
  - Barmherzige Bruder Krankenhaus Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Germany (2):
  - Charité Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Leipzig, Leipzig
- Hospital Universitario Quirónsalud Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 sites in 3 European countries. The first participant was enrolled on July 24, 2023 and the last participant had the last study visit on June 07,2024.
Pre-assignment Details: In this post-market study, the choice of BD Spinal NRFit™ needle (gauge, length, tip type), BD Syringes NRFit™, BD Spinal NRFit™ needle set, and BD Spinal Introducer NRFit™ needle was at clinician discretion. A total of 161 subjects were enrolled to ensure a minimum of 150 received spinal anesthesia and were observed for 10 days post-procedure for adverse events/complications. A minimum of 50 subjects per tip type (Quincke and Whitacre) were included.
Period: Overall Study
Arm/Group | All Participants
Started | 161
Enrolled Population (Participants who signed the informed consent) | 161
Treated Population (All participants in whom a spinal anesthesia procedure is attempted, regardless of success) | 153
Safety Population (All participants in whom a spinal anesthesia procedure is successful.) | 146
Completed | 153
Not Completed | 8
Not completed — Screen Failure | 2
Not completed — Withdrawal by Subject | 3
Not completed — Surgery cancelled | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All participants in whom a spinal anesthesia procedure is attempted, regardless of success.
Groups:
- Treated Population: Participants who underwent a neuraxial procedure, regardless of success.
Arm/Group | Treated Population
Number analyzed (Participants) | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (17.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 149
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  Austria | 59
  Germany | 49
  Spain | 45
Height [Mean (Standard Deviation); unit: cm] | 172.3 (9.47)
Weight [Mean (Standard Deviation); unit: Kg] | 80.76 (18.753)
Reasons for Surgery [Count of Participants; unit: Participants]
  Surgery of Lower Extremities | 91
  Surgery of Lower Abdomen | 40
  Surgery of Perineum | 4
  Surgery of Hips and Pelvis | 18
Reason for Neuraxial Procedure: Anesthesia [Count of Participants; unit: Participants] | 153
American Society of Anesthesiologists (ASA) Physical Status (PS) Classification [Count of Participants; unit: Participants] — The physician was responsible for assigning participants according to the ASA Physical Status classification:
  * ASA I: A normal healthy patient
  * ASA II: A patient with mild systemic disease
  * ASA III: A patient with severe systemic disease
  For a complete description, please refer to the study protocol.
  Participants
    I | 31
    II | 94
    III | 28
Participant position during spinal anesthesia [Count of Participants; unit: Participants]
  Lateral | 6
  Sitting | 147
Aseptic Technique [Count of Participants; unit: Participants]
  Chlorohexidine | 43
  Betadine | 10
  Octenidine | 32
  Other | 68
Local Anaesthesia [Count of Participants; unit: Participants]
  Lidocaine 1% | 113
  Lidocaine 2% | 35
  Other | 5
Number of Puncture Attempts [Count of Participants; unit: Participants]
  1 | 142
  2 | 10
  3 | 1
Lumbar interspace [Count of Participants; unit: Participants]
  L2-3 | 12
  L3-4 | 94
  L4-5 | 44
  Other | 3
Device Used [Count of Participants; unit: Participants]
  BD Spinal NRFit™ Needle Set | 128
  BD Spinal NRFit™ Needle | 25
BD Spinal NRFit™ Needle Type [Count of Participants; unit: Participants]
  BD Spinal NRFit™ Whitacre Needle | 103
  BD Spinal NRFit™ Quincke Needle | 50
Spontaneous appearance of CSF emerging from the needle hub [Count of Participants; unit: Participants] — Number of participants with a successful needle placement in the subarachnoid space defined as the appearance of cerebrospinal fluid (CSF) from the spinal needle hub
  Participants
    Spontaneous appearance of CSF emerging from the needle hub | 146
    No spontaneous appearance of CSF emerging from the needle hub | 7
BD NRFit™ Syringe Usage [Count of Participants; unit: Participants]
  BD Syringes NRFit™ Lok with a volume of 3 mL | 7
  BD Syringes NRFit™ Slip with a volume of 5 mL | 146
Ancillary device Usage [Count of Participants; unit: Participants]
  BD Blunt Fill NRFit™ Needle | 79
  BD Blunt Filter NRFit™ Needle | 74
Anesthetic medication aspiration [Count of Participants; unit: Participants]
  Anesthetic medication aspirated from vial | 43
  Anesthetic medication aspirated from ampule | 110
Anesthetic medication successfully aspirated using the BD NRFit™ syringe [Count of Participants; unit: Participants] | 153
Anesthetic medication injection through BD NRFit™ syringe [Count of Participants; unit: Participants]
  Anesthetic medication successfully injected through BD NRFit™ syringe | 146
  No anesthetic medication successfully injected through BD NRFit™ syringe | 7

OUTCOME MEASURES:

1. Primary Outcome: Primary Performance: Rate of Participants With Successful BD Spinal NRFit™ Needle Placement in the Subarachnoid Location
Description: Percentage of participants with successful placement of the BD Spinal NRFit™ needle in the subarachnoid location defined as the spontaneous appearance of cerebrospinal fluid (CSF) emerging from the spinal needle hub.
Time Frame: During insertion procedure
Population: All participants in whom a spinal anesthesia procedure is attempted, regardless of success.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 153
Participants
  Rate of successful placement of BD Spinal NRFit™ Whitacre Needle in subarachnoid location: number analyzed (Participants) | 103
  Rate of successful placement of BD Spinal NRFit™ Whitacre Needle in subarachnoid location | 100
  Rate of successful BD Spinal NRFit™ Quincke Needle placement in subarachnoid location: number analyzed (Participants) | 50
  Rate of successful BD Spinal NRFit™ Quincke Needle placement in subarachnoid location | 46
  Rate of successful BD Spinal NRFit™ Needle placement in subarachnoid location | 146

2. Primary Outcome: Primary Performance: Rate of of Participants With Successful Needle Placement in the Subarachnoid Location When a BD Spinal NRFit™ Introducer is Used
Description: Percentage of participants with successful placement of the BD Spinal NRFit™ needle in the subarachnoid location defined as the spontaneous appearance of cerebrospinal fluid (CSF) emerging from the spinal needle hub when an BD NRFit™ introducer is used.
Time Frame: During insertion procedure
Population: All participants in whom a spinal anesthesia procedure is attempted using a BD NRFit™ Spinal Introducer, regardless of success.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 130
Participants | 124

3. Primary Outcome: Primary Performance: Rate of Participants With Successful Aspiration Through BD NRFit™ Syringes
Description: Percentage of participants with successful aspiration of anesthetic through a BD NRFit™ Syringe.
Time Frame: During insertion procedure
Population: All participants in whom a spinal anesthesia procedure is attempted, regardless of success
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 153
Participants | 153

4. Primary Outcome: Primary Performance: Rate of Participants With BD NRFit™ Syringes That do Not Leak at the Connection Point During Medication Administration
Description: Percentage of participants with BD NRFit™ Syringes that do not leak at the connection point during medication administration.
Time Frame: During insertion procedure
Population: All participants in whom a spinal anesthesia procedure is successful
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 146
Participants | 145

5. Primary Outcome: Primary Safety: Rate of Participants With a Diagnosis of Post Dural Puncture Headache (PDPH)
Description: Percentage of participants with a diagnosis of PDPH (defined as headache that worsens when standing/upright position and relieves when laying supine) for a period of up to 10 (± 3 days) days following the procedure.
Time Frame: From insertion up to 10 (± 3 days) post procedure
Population: All participants in whom a spinal anesthesia procedure is successful
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 146
Participants
  Rate of post dural puncture headache (PDPH) for Subjects Using Whitacre Needle: number analyzed (Participants) | 100
  Rate of post dural puncture headache (PDPH) for Subjects Using Whitacre Needle | 1
  Rate of post dural puncture headache (PDPH) for Subjects Using Quincke Needle: number analyzed (Participants) | 46
  Rate of post dural puncture headache (PDPH) for Subjects Using Quincke Needle | 2
  Rate of post dural puncture headache (PDPH) | 3

6. Primary Outcome: Primary Safety: Percentage of Participants With Any Study Device and Procedure Adverse Events
Description: Percentage of participants with any device/procedure-related adverse events.
Time Frame: From insertion up to 10 (± 3 days) post procedure
Population: All participants in whom a spinal anesthesia procedure is attempted, regardless of success
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Population
Number analyzed (Participants) | 153
Participants
  Rate of participants with any BD NRFit™ spinal needle related adverse events (other than PDPH) | 0
  Rate of participants with any BD NRFit™ introducer-related adverse events (other than PDPH) | 0
  Rate of participants with any BD NRFit™ syringe-related adverse events (other than PDPH) | 0
  Rate of participants with any procedure-related adverse events (other than PDPH) | 6
  Rate of participants with any BD NRFit™spinal needle, introducer, syringe, or procedure-related AEs | 6

7. Primary Outcome: Primary Performance: Rate of of Participants With Successful Injection of Anesthetic Through BD NRFit™ Syringes
Description: Percentage of participants with successful injection of anesthetic through a BD NRFit™ Syringe.
Time Frame: During the insertion procedure
Population: All participants in whom a spinal anesthesia procedure is successful
Measure: Count of Participants; unit: Participants
Groups:
- Safety Population: All participants in whom a spinal anesthesia procedure is successful
Arm/Group | Safety Population
Number analyzed (Participants) | 146
Participants | 146

ADVERSE EVENTS:
Time Frame: From the spinal anesthesia up to 10 days (± 3 days) post procedure
Description: An Adverse Event is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, users, or other persons, whether or not related to the investigational medical devices or procedure and whether anticipated or unanticipated. Please refer to ISO 14155:2020 for serious adverse event definition.
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/153
Serious Adverse Events (participants affected / at risk) | 1/153
Other Adverse Events (participants affected / at risk) | 14/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=153)
Hypoaesthesia (Nervous system disorders) | 1 (1) — One SAE occurred in 1 of 153 subjects undergoing a neuraxial procedure. Due to prolonged hypesthesia possibly related to the spinal procedure, surgery could not be performed outpatient, requiring overnight hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=153)
Vertigo (Ear and labyrinth disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Urinary tract infection (Infections and infestations) | 1
Procedural headache (Injury, poisoning and procedural complications) | 3
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Presyncope (Nervous system disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT05953363/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT05953363/SAP_001.pdf